CLINICAL TRIAL: NCT00434902
Title: Evaluation of the Characteristics, Prevalence and Prognosis of Pulmonary Hypertension in Adult Patients With Sickle Cell Disease: Study ETENDARD.
Brief Title: Evaluation of the Prevalence of Pulmonary Hypertension in Adult Patients With Sickle Cell Disease
Acronym: ETENDARD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: PO51082; AOM-05037
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-11

CONDITIONS: Sickle Cell Disease
Keywords: Doppler Echocardiography; Pulmonary hypertension; Sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Recent data show that pulmonary hypertension (PH), defined by a tricuspid regurgitation jet (TRJ) velocity > or equal at 2.5m/s on Doppler echocardiography, is present in about 30% of adults with sickle cell disease (SCD) and is associated with poor prognosis. However in SCD the occurrence of PH (defined by mean pulmonary arterial pressure (mPAP)> or equal at 25 mmHg) is related to at least 3 mechanisms: PH due to hyperkinetic state with high cardiac output (CO) but normal pulmonary vascular resistance (PVR <160 dynes), or postcapillary PH (pulmonary capillary wedge pressure PCWP >15 mmHg), or precapillary pulmonary arterial hypertension (PAH) defined by mPAP > or equal at 25 mmHg, PCWP< or equal at 15 mmHg and PVR > or equal at 160 dynes.The aim of this study is to evaluate in a French population of adults with sickle cell disease the characteristics, prevalence and prognosis of pulmonary hypertension.

DETAILED DESCRIPTION:
Consecutive adult patients with sickle cell disease (SCD) had a Doppler echocardiography to evaluate if they had a suspected pulmonary hypertension (PH) on the basis of a tricuspid regurgitation jet (TRJ) velocity > or equal at 2.5m/s. In this case, a right heart catheterization was performed to confirm or not this diagnosis and its mechanisms. Each included patient was followed every year for 3 years: during each visit, a clinical evaluation was obtained and a Doppler echocardiography. In case of emergence of a suspected PH, a right heart catheterization was performed to confirm or not this diagnosis and its mechanisms.

Three groups of patients were defined: no PH, precapillary PH, and a third group including post-capillary PH and hyperkinetic state. These groups were well defined on the basis of the results of th Doppler echocardiography and right heart catheterisation.

Characteristics of patients and their prognosis were evaluated in each group.

In the same, way, biological study is planned to evaluate some biological markers of the mechanism of PH, and prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous SS sickle cell disease
* Male or female > 18 years of age
* VOC (Vaso-Occlusive crisis) or ACS (Acute chest syndrome)within 6 weeks of inclusion ("Stable state")
* Signed written Informed consent

Exclusion Criteria:

* Creatinine clearance < 30 ml/mn
* prothrombin ratio < 50%
* Severe pneumopathy and TLC (Total lung capacity) < 70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients With Sickle Cell Disease
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-03 (Actual); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald SIMONNEAU, MD, Principal Investigator — Hôpital Antoine Béclère, CLAMART; Frederic Galacteros, MD, Principal Investigator — Hôpital Henri Mondor, Creteil; Serge ADNOT, MD, Study Director — Hôpital Henri Mondor, CRETEIL; Bernard MAITRE, MD, Study Director — Hopital Henri Mondor, CRETEIL; Marc HUMBERT, MD, Study Director — Hôpîtal Antoine Béclere, CLAMART; Robert GIROT, MD, Study Director — Hôpital Tenon, PARIS; François LIONNET, MD, Study Director — Hôpital TENON, PARIS; Françoise DRISS, MD, Study Director — Hôpital Bicêtre, KREMLIN BICETRE; Olivier LAMBOTTE, MD, Study Chair — Hôpital Bicêtre, KREMLIN BICETRE; Jocelyn INAMO, MD, Study Director — CHU Fort de France; Gylna LOKO, MD, Study Director — CHU Fort de France; Olivier SITBON, MD, Study Director — Hôpital Antoine Béclère, CLAMART; Xavier Jaïs, MD, Study Director — Hôpital Antoine Béclère, CLAMART; Anoosha Habibi, MD, Study Chair — Hôpital Henri Mondor, CRETEIL; Dora Bachir, MD, Study Chair — Hôpital Henri Mondor, CRETEIL; Laurent SAVALE, MD, Study Chair — Hopital Henri Mondor, CRETEIL; Saadia Eddahibi, MD, Study Chair — Hôpital Henri Mondor, CRETEIL; Gilles Garcia, MD, Study Chair — Hopital Antoine Béclère, CLAMART
Locations (1):
- Hôpital Antoine Béclère, Clamart, France

REFERENCES:
- [Background] Simonneau G, Galie N, Rubin LJ, Langleben D, Seeger W, Domenighetti G, Gibbs S, Lebrec D, Speich R, Beghetti M, Rich S, Fishman A. Clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2004 Jun 16;43(12 Suppl S):5S-12S. doi: 10.1016/j.jacc.2004.02.037. PMID 15194173
- [Background] Rubin LJ, Badesch DB, Barst RJ, Galie N, Black CM, Keogh A, Pulido T, Frost A, Roux S, Leconte I, Landzberg M, Simonneau G. Bosentan therapy for pulmonary arterial hypertension. N Engl J Med. 2002 Mar 21;346(12):896-903. doi: 10.1056/NEJMoa012212. PMID 11907289
- [Background] Humbert M, Sitbon O, Simonneau G. Treatment of pulmonary arterial hypertension. N Engl J Med. 2004 Sep 30;351(14):1425-36. doi: 10.1056/NEJMra040291. No abstract available. PMID 15459304
- [Background] Lechapt E, Habibi A, Bachir D, Galacteros F, Schaeffer A, Desvaux D, Brochard L, Housset B, Godeau B, Maitre B. Induced sputum versus bronchoalveolar lavage during acute chest syndrome in sickle cell disease. Am J Respir Crit Care Med. 2003 Dec 1;168(11):1373-7. doi: 10.1164/rccm.200302-174OC. Epub 2003 Sep 11. PMID 12969866
- [Background] Maitre B, Habibi A, Roudot-Thoraval F, Bachir D, Belghiti DD, Galacteros F, Godeau B. Acute chest syndrome in adults with sickle cell disease. Chest. 2000 May;117(5):1386-92. doi: 10.1378/chest.117.5.1386. PMID 10807826
- [Derived] Simon T, Savale L, Grundtvig Skaarup K, Breillat P, Pham LL, Nouraie SM, Dyrby Johansen N, Inamo J, Lionnet F, Loko G, Chantalat C, Pham Hung d'Alexandry d'Orengiani AL, Habibi A, de Luna G, Iles S, Galacteros F, Audureau E, Biering-Sorensen T, Bartolucci P, Derumeaux G, d'Humieres T. Sickle Cell Diastolic Cardiomyopathy and Mortality Risk: A Novel Echocardiographic Framework for Prognostic Stratification. Am J Hematol. 2025 Nov;100(11):1940-1951. doi: 10.1002/ajh.27768. Epub 2025 Jul 22. PMID 40693500
- [Derived] Parent F, Bachir D, Inamo J, Lionnet F, Driss F, Loko G, Habibi A, Bennani S, Savale L, Adnot S, Maitre B, Yaici A, Hajji L, O'Callaghan DS, Clerson P, Girot R, Galacteros F, Simonneau G. A hemodynamic study of pulmonary hypertension in sickle cell disease. N Engl J Med. 2011 Jul 7;365(1):44-53. doi: 10.1056/NEJMoa1005565. PMID 21732836